CLINICAL TRIAL: NCT02357160
Title: The Value of Integrating Visual Arts (VIVA): Evaluating the Benefits of Hospital Room Artwork on Inpatient Wellbeing
Brief Title: The Value of Integrating Visual Arts: Evaluating the Benefits of Hospital Room Artwork on Inpatient Wellbeing
Acronym: VIVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Daniel R George, Assistant Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00000378
Record Dates: First submitted 2015-01-29; First posted 2015-02-06 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Choice (Experimental): Patients given choice over artwork on wall
  Interventions: Behavioral: Artwork
- No choice (Active Comparator): Patients not given choice over artwork on wall
  Interventions: Behavioral: Artwork
- No artwork (Placebo Comparator): Patients not receiving any artwork on wall
  Interventions: Behavioral: Artwork

INTERVENTIONS:
Behavioral: Artwork — Prints by local artists that are hung on the walls of patient rooms.

SUMMARY:
The Value of Integrating Visual Arts (VIVA): Evaluating the Benefits of Hospital Room Artwork on Inpatient Wellbeing will use a large randomized controlled trial design to investigate how the inclusion of visual arts in the hospital rooms of cancer patients benefits their quality-of-life during treatment. This 18-month research study will provide hospitals with evidence of the therapeutic value of the visual arts as measured by patients' perceptions of anxiety, pain ratings, use of pain medications, need for nurses, and length of stay. Data also will be collected on patients' evaluation of hospital rooms, specifically on décor including artwork, so as to correlate patient wellbeing with the presence of artwork. Ultimately, this project aims to increase support of and appreciation for the arts from a major consumer-namely, healthcare providers-by justifying the value of integrating local visual art into inpatient rooms and providing patients with aesthetic choice during their stay.

DETAILED DESCRIPTION:
The arts have long played a role in health and healing dating back to the 14th century when paintings ushered patients to a good death or immortalized patrons for charitable activities. Today, about half of all hospitals have dedicated art programs ranging from permanent displays of art throughout their buildings to art therapies at the bedside and performances in public spaces such as waiting areas. Offered to patients with a range of conditions, their families and visitors, those programs aim to "improve patients' overall health outcomes, treatment compliance and quality of life". Yet, while patient surveys indicate interior design features such as artwork can make hospital environments less institutionalized and more emotionally pleasing, few randomized controlled trials have linked specific design features or interventions directly to impacts on healthcare outcomes. The Value of Integrating Visual Arts: Evaluating the Benefits of Hospital Room Artwork on Inpatient Wellbeing will add significantly to those data.

The physical environment of the inpatient hospital room essentially provides a blank canvas on which to study the impact of visual arts on patient outcomes. Studies show that patients care about their physical surroundings, and while efforts in recent years have aimed to make hospital rooms less austere, in most cases, they remain institutional environments. The Pick-a-Pic Program at the Penn State Milton S. Hershey Medical Center addresses this problem by allowing patients to modify one aspect of their physical environment through the personal selection of an art print by a local, professional artist to be displayed in their rooms during their hospitalization. Placed in frames mounted on the walls directly in patients' line of vision from their hospital beds, these prints can help to create a supportive and comforting environment. Their efficacy is predicated on the capacity of visual arts to provide positive distractions for patients and family members coping with the stress of illness by adding a personal touch to the hospital environment and making the spaces as familiar and homelike as possible.

This project draws upon distraction theory, which posits that patients who become engrossed in or open to a positive distraction attend less to their pain and even experience reduced or altered perceptions of pain. Changing even one environmental factor-such as introducing a visual stimulus-can provide that distraction. Burn patients, for instance, who watch videos of nature scenes with accompanying music during burn dressing changes were found to experience less pain and report less anxiety. Similar findings were reported for those patients who viewed a nature scene and heard nature sounds while undergoing a painful flexible bronchoscopy. In studies involving healthy volunteers, participants shown videos of nature scenes-some with music and some without-had higher pain thresholds and pain tolerance than volunteers who stared at blank or black screens. Positive distractions as part of the healthcare physical environment also have been found to be effective in diminishing feelings of stress and its accompanying psychological and physiological impacts. When videos, still art, and window film of nature images were introduced into two emergency departments, researchers noted reductions in behaviors indicative of stress and anxiety. Artwork has been found to have a positive effect on patients' moods as well.

The proposed study - The Value of Integrating Visual Arts (VIVA): Evaluating the Benefits of Hospital Room Artwork on Inpatient Wellbeing - builds on these findings and advances them in novel and significant ways. First, this is a rare three-arm randomized controlled trial with large participant numbers designed to quantitatively assess the benefit of visual arts to individuals. The participants in our study represent a specific subgroup-i.e., patients-with a discrete disease diagnosis of cancer who are undergoing treatment in the Cancer Institute at the Penn State Hershey Medical Center. According to the Center for Disease Control, more than 19 million adults, or almost one in ten Americans, have been diagnosed with cancer. Widely known as one of the most disruptive illnesses affecting human beings, cancer treatment is painful and invasive, and patients and their families must cope with feelings of anxiety, vulnerability, and uncertainty - feelings that can be exacerbated by the stark medicalized environment. Positive visual stimulus in the form of artwork has the capacity to provide biopsychosocial respite that can be captured in measurable patient outcomes from this physical and psychological trauma. While this research study is particularly relevant for cancer patients, findings of this project holds promise for all hospital inpatients who are subject to the same sorts of environmental stimuli as they undergo institutional treatment. According to the CDC, there are a reported 35.1 million inpatients annually receiving care in U.S. hospitals, and the average length of stay is 4.8 days. As clinical and economic data have traditionally carried the greatest weight in decisions by hospital administrators, this study has the potential to produce strong scientific data establishing the visual arts as an environmental modification with clear and persuasive benefits for a hospital and its patients that deserves investment.

This study also is innovative in linking measurable patient outcomes to patient control of one aspect of the hospital physical environment-namely, artwork for inpatient rooms. Studies that have examined artwork and physiological outcomes have largely involved views of nature from windows or representational nature scenes, both of which have been provided to rather than chosen by patients. In studies involving patient choice, the focus often has been to determine patients' preferences for different kinds of artwork-e.g., representational nature scenes vs. abstract, rural scenes vs. urban-with an eye to developing guidelines for art selection and placement. While qualitative data exist that show patients who are able to influence their physical environment report increased feelings of emotional and physical comfort as well as improved moods, few studies have used rigorous study designs to measure the benefit of choice of artwork on medical outcomes.

Finally, this study is innovative in using a single lens-visual arts-to examine the benefits of the arts in hospital rooms on patient satisfaction, a key parameter to healthcare providers in today's competitive market. Other examinations of the physical environment have included architectural features such as size and shape of hospital rooms, ambient features such as lighting and temperature, and colors. By specifying room décor in patient satisfaction surveys, this study can provide hospitals with strong and persuasive data on a relatively low-cost way to improve the aesthetics of patients' rooms. Indeed, prints of artwork used in the Pick-a-Pic program at the medical center cost about $90 to produce.

This research study seeks to answer (1) whether the presence of visual arts in a patient's hospital room significantly improves patient outcomes as measured by perceptions of anxiety, reports of pain, use of pain medications, requests for nursing staff; (2) whether patient's personal choice of a visual arts print (versus having a print but no choice) significantly improves those outcomes; and (3) whether the presence of visual arts significantly improves patient satisfaction with the physical environment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are admitted to the Penn State Hershey Cancer Institute (7th floor) for treatments including oncology, bone marrow transplant, and hematology. Patients will be 18 years or older

Exclusion Criteria:

* Patients whose treatments do not include oncology, bone marrow transplant, and hematology; who are not hospitalized on the 7th floor of the Cancer Institute; and who are not 18 years or older.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Perceptions of anxiety as measured by the State-Trait Anxiety Inventory for Adults | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks

SECONDARY OUTCOMES:
Reports of pain as drawn for each patient via PowerChart, the hospital's electronic medical record software for documenting patient care | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Use of pain medications as drawn for each patient via PowerChart, the hospital's electronic medical record software for documenting patient care | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Mood as measured by the Mitchell Emotional Thermometer | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel George, PhD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] George DR, Boer C, Hammer J, Hopkins M, King T, Green MJ. Evaluating the Benefits of Hospital Room Artwork for Patients Receiving Cancer Treatment: A Randomized Controlled Trial. J Hosp Med. 2018 Aug 1;13(8):558-561. doi: 10.12788/jhm.2915. Epub 2018 Feb 5. PMID 29401210